CLINICAL TRIAL: NCT00447395
Title: Genetic Abnormalities and Oxidative Stress in Sperm as Cause of Recurrent Miscarriage.
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Jose Bellver, Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: VLC-JB-1106-307-4
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Recurrent Miscarriage
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- GROUP 1: Recurrent miscarriage, <40 year-old-men, < 38 year-old-women, normal or mild affected sperm, normal parents karyotype, no thrombophilia, normal uterus, no endocrinopathy
- GROUP 2: •Recurrent miscarriage, <40 year-old-men, < 38 year-old-women, oligozoospermia (1-5 mill/ml), normal parents karyotype, no thrombophilia, normal uterus, no endocrinopathy
- GROUP 3: •Oligozoospermia (1-5 mill/ml), < 40 year-old-men, no recurrent miscarriages
- GROUP 4: •Healthy young sperm donors

SUMMARY:
In recurrent miscarriage, the male factor has been poorly evaluated. In fact, in the vast majority of clinical protocols of recurrent miscarriage, the sperm is not considered or assessed. Recently, some studies have suggested the presence of genetic and metabolic sperm anomalies in couples suffering from repeated miscarriages. Specifically, DNA fragmentation and altered oxidative stress in the sperm and Y microdeletions from blood samples have been related to an increased risk of miscarriage.The aim of the present study is to compare these three parameters in: couples with recurrent miscarriage; oligozoospermic men with or without recurrent miscarriages; and healthy sperm donors, in order to determine their actual impact on this reproductive problem.

ELIGIBILITY:
Inclusion Criteria:

4 groups

* Recurrent miscarriage, <40 year-old-men, < 38 year-old-women, normal or mild affected sperm, normal parents karyotype, no thrombophilia, normal uterus, no endocrinopathy
* The same criteria than in group A, but oligozoospermia (1-5 mill/ml)
* Oligozoospermia (1-5 mill/ml), < 40 year-old-men, no recurrent miscarriages
* Healthy young sperm donors

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples with recurrent miscarriages
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Bellver, MD, Principal Investigator — IVI Valencia
Locations (1):
- Ivi Valencia, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Bellver J, Meseguer M, Muriel L, Garcia-Herrero S, Barreto MA, Garda AL, Remohi J, Pellicer A, Garrido N. Y chromosome microdeletions, sperm DNA fragmentation and sperm oxidative stress as causes of recurrent spontaneous abortion of unknown etiology. Hum Reprod. 2010 Jul;25(7):1713-21. doi: 10.1093/humrep/deq098. Epub 2010 May 24. PMID 20501469